CLINICAL TRIAL: NCT01892657
Title: Cetaphil® Daily Facial Moisturizer With Sunscreen SPF 50+ - Human Repeat Insult Patch Test Skin Irritation/Sensitization Evaluation (Semi-occlusive Patch)
Brief Title: Cetaphil® Daily Facial Moisturizer With Sunscreen SPF 50+ - Human Repeat Insult Patch Test
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GLI.04.SRE.US10093
Record Dates: First submitted 2013-07-01; First posted 2013-07-04 (Estimated); Results first posted 2013-09-25 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2008-08

CONDITIONS: Skin Irritation
Keywords: Cetaphil Daily Facial Moisturizer with SPF 50+; Hypoallergenicity; Skin Irritation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Facial Moisturizer with SPF 50+ (Experimental): All subjects received Cetaphil Daily Facial Moisturizer with SPF 50+
  Interventions: Drug: Facial Moisturizer with SPF 50+

INTERVENTIONS:
Drug: Facial Moisturizer with SPF 50+ — All subjects received applications of occlusive patches dosed with Cetaphil Daily Facial Moisturizer with SPF 50+
  Other Names: Cetaphil Daily Facial Moisturizer with SPF 50+

SUMMARY:
This study examined the possible sensitization and irritation effects of a moisturizer with sunscreen SPF 50+.

DETAILED DESCRIPTION:
The design for this study is standard for human repeat insult patch tests. To test the moisturizer with sunscreen SPF 50+ for the potential to induce contact sensitization by repetitive applications, healthy subjects received 9 applications at 48 to 72 hour intervals of the moisturizer to the upper back. Patches were remained on the skin for approximately 48 to 72 hours. Twelve to 24 days after the previous applications, subjects were patched with the moisturizer at the original site and an alternative site for 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 to 70 years of age in general good health
* Can read, understand, and sign informed consent

Exclusion Criteria:

* History of acute or chronic disease
* Diagnosed with chronic skin allergies
* Pregnant or lactating

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Gottschalk, MD, Study Director — Galderma R&D
Locations (1):
- Thomas J. Stephens and Associates, Inc., Colorado Springs, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened at a single US center.
Period: Overall Study
Arm/Group | Facial Moisturizer With SPF 50+
Started | 128
Completed | 110
Not Completed | 18
Not completed — Withdrawal by Subject | 6
Not completed — Protocol Violation | 12

BASELINE CHARACTERISTICS:
Population: All subjects who were enrolled in the study and participated in all scheduled visits during the study were analyzed.
Arm/Group | Facial Moisturizer With SPF 50+
Number analyzed (Participants) | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 109
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (13.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86
  Male | 24
Race/Ethnicity, Customized [Number; unit: Participants]
  African American | 10
  Asian | 3
  Caucasian | 71
  Hispanic | 23
  Caucasian/Hispanic | 3
Region of Enrollment [Number; unit: participants]
  United States | 110

OUTCOME MEASURES:

1. Primary Outcome: Area of Erythema and Elevated Responses of Skin to Product
Description: Subjects were patched 9 times at 48 hour to 72 hour intervals and graded for erythema and elevated responses (edema, papules, vesicles, bullae) on a 4 point scale (0 = none, 1 = mild, 2 = moderate, 3 = severe). 12 to 24 hours after the last patch application, a challenge patch was applied at the same site and a challenge patch was applied to an alternate site. Both were graded for the same criteria at 48 hours and at 96 hours. A total of 11 patches were applied to each subject. All patches were removed after 48 hours.
Time Frame: 3 consecutive weeks
Measure: Number; unit: participants
Groups:
- Patch 1; Patch 2; Patch 3; Patch 4; Patch 5; Patch 6; Patch 7; Patch 8; Patch 9: Subjects received a patch dosed with 100 microliters of Cetaphil Daily Facial Moisturizer with SPF 50+
- Challenge Patch (Original Site) - 48 Hours: The challenge patch dosed with 100 microliters of Cetaphil Daily Facial Moisturizer with SPF 50+ applied to the original application site was graded at 48 hours.
- Challenge Patch (Original Site) - 96 Hours: The challenge patch dosed with 100 microliters of Cetaphil Daily Facial Moisturizer with SPF 50+ applied to the original application site was graded again at 96 hours.
- Challenge Patch (Alternate Site) - 48 Hours: A challenge patch dosed with 100 microliters of Cetaphil Daily Facial Moisturizer with SPF 50+ applied to an alternate application site was graded at 48 hours.
- Challenge Patch (Alternate Site) - 96 Hours: A challenge patch dosed with 100 microliters of Cetaphil Daily Facial Moisturizer with SPF 50+ applied to an alternate application site was graded again at 96 hours.
Arm/Group | Patch 1 | Patch 2 | Patch 3 | Patch 4 | Patch 5 | Patch 6 | Patch 7 | Patch 8 | Patch 9 | Challenge Patch (Original Site) - 48 Hours | Challenge Patch (Original Site) - 96 Hours | Challenge Patch (Alternate Site) - 48 Hours | Challenge Patch (Alternate Site) - 96 Hours
Number analyzed (Participants) | 110 | 110 | 110 | 110 | 110 | 110 | 110 | 110 | 110 | 110 | 110 | 110 | 110
participants
  None | 91 | 68 | 33 | 42 | 39 | 20 | 33 | 33 | 23 | 78 | 85 | 86 | 95
  Mild | 19 | 41 | 72 | 68 | 69 | 82 | 72 | 72 | 78 | 31 | 24 | 23 | 12
  Moderate | 0 | 1 | 5 | 0 | 2 | 8 | 5 | 5 | 9 | 1 | 1 | 1 | 3

ADVERSE EVENTS:
Arm/Group | Facial Moisturizer With SPF 50+
Serious Adverse Events (participants affected / at risk) | 0/110
Other Adverse Events (participants affected / at risk) | 0/110

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less